CLINICAL TRIAL: NCT04786392
Title: Lutein Absorption Consumed as Supplement, Blended Food, or Wholefood Over 24-hours.
Brief Title: Food or Supplemental Lutein Absorption
Acronym: FSLA20
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to fit within PhD timeline.
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2020002809
Record Dates: First submitted 2021-02-26; First posted 2021-03-08 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-01

CONDITIONS: Macula Lutea Opacity
Keywords: lutein; absorption; supplement
MeSH Terms: interventions — Food; Airway Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lutein supplement (Active Comparator): Supplement containing 5 mg powdered lutein, capsule filler microcrystalline cellulose.
  To be administered once.
  Interventions: Dietary Supplement: Lutein supplement
- Blended food beverage (Experimental): Blended food beverage containing 5 mg lutein from baby spinach. To be administered/consumed once.
  Interventions: Other: Food, blended
- Whole food (Experimental): Consumption of 5 mg of lutein from baby spinach. To be administered/consumed once.
  Interventions: Other: Food, unprocessed

INTERVENTIONS:
Dietary Supplement: Lutein supplement — 5 mg lutein supplement.
  Arms: Lutein supplement
Other: Food, blended — 5 mg lutein from baby spinach, blended.
  Arms: Blended food beverage
Other: Food, unprocessed — 5 mg lutein from baby spinach, in whole food form.
  Arms: Whole food

SUMMARY:
The aim of this study is to investigate in healthy adults, 18-40 years of age, how the absorption of 5 mg of L differs between consumption as a supplement, blended foods, and whole food equivalent of blended foods.

DETAILED DESCRIPTION:
The absorption the macular carotenoids has shown variability between different supplements, and food sources such as egg and spinach. Investigation of the absorption of different forms of food (e.g. cooked, raw, blended) is not as well studied. Investigating the absorption of lutein from different forms of food is important to be able to prescribe lutein from forms of food that will be optimally absorbed.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 to 40 years.
* Generally healthy.
* No participant reported history of clinically significant medical conditions including, but not limited to, cardiovascular, neurological, psychiatric, renal, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled.
* Non-smoker.
* English language proficiency

Exclusion Criteria:

* Participant reported diagnosis of serious ocular conditions (e.g. cataracts, glaucoma, diabetic retinopathy, retinitis pigmentosa, Stagardt's disease)
* Participant reported diagnosis, or current treatment of age-related macular degeneration.
* Participant reported diagnosis of epilepsy.
* Participant aversion, intolerance or allergy to study foods to be consumed (spinach, ginger, lemon, apple, flaxseeds)
* A female currently pregnant or trying to fall pregnant.
* Current or past smoker (within last 12 months).
* Under 18 or over 40 years of age.
* Currently taking a lutein supplement or consuming large amounts of foods containing lutein on a regular basis (>3 days per week).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Plasma lutein concentration | Study visit 1 (24 hours), Study visit 2 (24 hours), study visit 3 (24 hours)
  Area under the curve of plasma lutein concentrations between 0 and 24 hours post lutein consumption.

SECONDARY OUTCOMES:
Plasma lutein maximum concentration | Study visit 1 (24 hours), Study visit 2 (24 hours), study visit 3 (24 hours)
  Maximum concentration of plasma lutein reached over 24 hours of measurement, and time point of maximum concentration.
Macular pigment optical density | Study visit day 1, day 8, day 15
  Machine: measured by the Macular Pigment Screener II (Elektron Eye Technology). The non-invasive test uses heterochromatic flicker photometry. One measure completed at each study visit (3 study visits total).
Daily dietary lutein and zeaxanthin intake | Study visit day 1
  Daily dietary intake of lutein and zeaxanthin (mg/day) as measured by a food frequency questionnaire.
Daily dietary lutein and zeaxanthin intake | Study visit day 1, day 8, day 15
  Daily dietary intake of lutein and zeaxanthin (mg/day) as measured by a food frequency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Chahay, PhD, Principal Investigator — The University of Queensland
Locations (1):
- School of Human Movement and Nutrition Sciences, The University of Queensland, Saint Lucia, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein PS, Li B, Vachali PP, Gorusupudi A, Shyam R, Henriksen BS, Nolan JM. Lutein, zeaxanthin, and meso-zeaxanthin: The basic and clinical science underlying carotenoid-based nutritional interventions against ocular disease. Prog Retin Eye Res. 2016 Jan;50:34-66. doi: 10.1016/j.preteyeres.2015.10.003. Epub 2015 Nov 2. PMID 26541886
- [Background] Chiu CJ, Chang ML, Zhang FF, Li T, Gensler G, Schleicher M, Taylor A. The relationship of major American dietary patterns to age-related macular degeneration. Am J Ophthalmol. 2014 Jul;158(1):118-127.e1. doi: 10.1016/j.ajo.2014.04.016. Epub 2014 Apr 29. PMID 24792100
- [Background] Wu J, Seregard S, Algvere PV. Photochemical damage of the retina. Surv Ophthalmol. 2006 Sep-Oct;51(5):461-81. doi: 10.1016/j.survophthal.2006.06.009. PMID 16950247
- [Background] Widomska J, Subczynski WK. Why has Nature Chosen Lutein and Zeaxanthin to Protect the Retina? J Clin Exp Ophthalmol. 2014 Feb 21;5(1):326. doi: 10.4172/2155-9570.1000326. PMID 24883226
- [Background] Liu T, Liu WH, Zhao JS, Meng FZ, Wang H. Lutein protects against beta-amyloid peptide-induced oxidative stress in cerebrovascular endothelial cells through modulation of Nrf-2 and NF-kappab. Cell Biol Toxicol. 2017 Feb;33(1):57-67. doi: 10.1007/s10565-016-9360-y. Epub 2016 Nov 22. PMID 27878403
- [Background] Frede K, Ebert F, Kipp AP, Schwerdtle T, Baldermann S. Lutein Activates the Transcription Factor Nrf2 in Human Retinal Pigment Epithelial Cells. J Agric Food Chem. 2017 Jul 26;65(29):5944-5952. doi: 10.1021/acs.jafc.7b01929. Epub 2017 Jul 13. PMID 28665123
- [Background] Howells O, Eperjesi F, Bartlett H. Measuring macular pigment optical density in vivo: a review of techniques. Graefes Arch Clin Exp Ophthalmol. 2011 Mar;249(3):315-47. doi: 10.1007/s00417-010-1577-5. Epub 2011 Jan 8. PMID 21221629
- [Background] Kopsell DA, Lefsrud MG, Kopsell DE, Wenzel AJ, Gerweck C, Curran-Celentano J. Spinach cultigen variation for tissue carotenoid concentrations influences human serum carotenoid levels and macular pigment optical density following a 12-week dietary intervention. J Agric Food Chem. 2006 Oct 18;54(21):7998-8005. doi: 10.1021/jf0614802. PMID 17032001
- [Background] van der Made SM, Kelly ER, Kijlstra A, Plat J, Berendschot TT. Increased Macular Pigment Optical Density and Visual Acuity following Consumption of a Buttermilk Drink Containing Lutein-Enriched Egg Yolks: A Randomized, Double-Blind, Placebo-Controlled Trial. J Ophthalmol. 2016;2016:9035745. doi: 10.1155/2016/9035745. Epub 2016 Mar 14. PMID 27064326
- [Background] Taibi G, Nicotra CM. Development and validation of a fast and sensitive chromatographic assay for all-trans-retinol and tocopherols in human serum and plasma using liquid-liquid extraction. J Chromatogr B Analyt Technol Biomed Life Sci. 2002 Nov 25;780(2):261-7. doi: 10.1016/s1570-0232(02)00529-9. PMID 12401351
- [Background] Chung HY, Rasmussen HM, Johnson EJ. Lutein bioavailability is higher from lutein-enriched eggs than from supplements and spinach in men. J Nutr. 2004 Aug;134(8):1887-93. doi: 10.1093/jn/134.8.1887. PMID 15284371
- [Background] Aebischer CP, Schierle J, Schuep W. Simultaneous determination of retinol, tocopherols, carotene, lycopene, and xanthophylls in plasma by means of reversed-phase high-performance liquid chromatography. Methods Enzymol. 1999;299:348-62. doi: 10.1016/s0076-6879(99)99035-3. No abstract available. PMID 9916214